CLINICAL TRIAL: NCT00017004
Title: Phase III Trial to Evaluate the Efficacy of Maintaining Hemoglobin Levels Above 120 g/l With Erythropoietin Versus Above 100 g/l Without Erythropoietin in Anemic Patients Receiving Concurrent Radiation and Cisplatin for Cervical Cancer
Brief Title: Radiation Therapy and Cisplatin With or Without Epoetin Alfa in Treating Patients With Cervical Cancer and Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: Canadian Cancer Trials Group (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GOG-0191; NCI-2012-02384 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CAN-NCIC-CX4; CDR0000068641; GOG-0191 (Other: Gynecologic Oncology Group); GOG-0191 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Anemia; Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma; Drug Toxicity; Radiation Toxicity; Stage IIB Cervical Cancer; Stage III Cervical Cancer; Stage IVA Cervical Cancer
MeSH Terms: conditions — Anemia; Drug-Related Side Effects and Adverse Reactions; Radiation Injuries; Uterine Cervical Neoplasms | interventions — Cisplatin; Brachytherapy; Epoetin Alfa; Erythropoietin

ARMS (2):
- Arm I (Experimental): Patients undergo radiotherapy comprising pelvic external beam radiotherapy daily five days a week for 5 weeks, followed by either 1 or 2 implants of low-dose rate intracavitary brachytherapy or 5 fractions of high-dose rate intracavitary brachytherapy, followed by 3-5 days of parametrial boost radiotherapy. Patients receive cisplatin IV concurrently with pelvic external beam radiotherapy on days 1, 8, 15, 22, 29, and once during the week of parametrial boost radiotherapy.
  Interventions: Radiation: External Beam Radiation Therapy; Drug: Cisplatin; Radiation: Internal Radiation Therapy
- Arm II (Experimental): Patients undergo radiotherapy and chemotherapy as in arm I. Additionally, patients receive epoetin alfa subcutaneously once weekly concurrently with radiotherapy and chemotherapy.
  Interventions: Radiation: External Beam Radiation Therapy; Drug: Cisplatin; Radiation: Internal Radiation Therapy; Biological: Epoetin Alfa

INTERVENTIONS:
Radiation: External Beam Radiation Therapy — Undergo radiation
  Other Names: Definitive Radiation Therapy; EBRT; External Beam RT
Drug: Cisplatin — Given IV
Radiation: Internal Radiation Therapy — Undergo radiation
  Other Names: Brachytherapy; Internal Radiation; Internal Radiation Brachytherapy; Radiation Brachytherapy
Biological: Epoetin Alfa — Given SC
  Other Names: EPO; Epogen; Eprex; erythropoietin; r-HuEPO
  Arms: Arm II

SUMMARY:
Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Epoetin alfa may stimulate red blood cell production to treat anemia in patients who have received chemotherapy and/or radiation therapy for cervical cancer. Randomized phase III trial to study the effectiveness of epoetin alfa in treating anemia in patients who have cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Assess the efficacy of raising and maintaining hemoglobin (Hgb) levels above 12.0 g/dL with epoetin alfa vs maintaining Hgb levels above 10.0 g/dL without epoetin alfa on progression-free survival, overall survival, and local control in anemic patients with cervical cancer receiving concurrent radiotherapy and cisplatin. Compare the quality of life of patients treated with these regimens.

OUTLINE:

This is a randomized study. Patients are stratified according to stage (IIB vs IIIB vs IVA), method of brachytherapy (low-dose vs high-dose), and surgical staging of para-aortic nodes (yes vs no). Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients undergo radiotherapy comprising pelvic external beam radiotherapy daily five days a week for 5 weeks, followed by either 1 or 2 implants of low-dose rate intracavitary brachytherapy or 5 fractions of high-dose rate intracavitary brachytherapy, followed by 3-5 days of parametrial boost radiotherapy. Patients receive cisplatin IV concurrently with pelvic external beam radiotherapy on days 1, 8, 15, 22, 29, and once during the week of parametrial boost radiotherapy.

Arm II: Patients undergo radiotherapy and chemotherapy as in arm I. Additionally, patients receive epoetin alfa subcutaneously once weekly concurrently with radiotherapy and chemotherapy. Quality of life is assessed at baseline, during weeks 3 and 6, within 1 week of last brachytherapy, and every 3 months for 2 years. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 460 patients will be accrued for this study within 3.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the cervix

  * Stage IIB, IIIB, or IVA
  * Primary, previously untreated disease
* Hemoglobin less than 14 g/dL at presentation
* Negative, non-suspicious para-aortic nodes determined by lymphangiogram, CT scan, MRI, or lymphadenectomy
* Eligible for treatment with radical intent involving concurrent cisplatin and pelvic radiotherapy
* No involvement of the lower third of vagina
* No carcinoma of the cervical stump
* Performance status - GOG 0-3
* See Disease Characteristics
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 3 times normal
* Alkaline phosphatase no greater than 3 times normal
* Creatinine no greater than 2.0 mg/dL
* No uncontrolled hypertension
* No history of thrombotic vascular events (e.g., deep vein thrombosis or myocardial infarction)
* No active hemolysis
* No history of pulmonary embolism
* No septicemia or severe infection
* No circumstances that would preclude study participation
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No history of hypersensitivity to epoetin alfa or human albumin
* No diagnosis of vitamin B_12 or folic acid deficiency
* No recent (within the past 3 months) or uncontrolled seizure disorder
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* See Disease Characteristics
* See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2001-08; Primary Completion 2004-05-15 (Actual)

PRIMARY OUTCOMES:
Progression-free survival with progression defined as a 50% or greater increase in the cross-product of the existing primary tumor relative to the smallest cross-product from all previous exams | Up to 5 years

SECONDARY OUTCOMES:
Overall survival | Up to 5 years
Local control, coded as successful if any relapse or disease progression is is contained within the pelvic field | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Thomas, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group of Arizona, Phoenix, Arizona, United States